CLINICAL TRIAL: NCT02036112
Title: Randomized Clinical Trial of Conventional Versus Individual Extralevator Abdominoperineal Excision for Locally Advanced Lower Rectal Cancer
Brief Title: Conventional Versus Individual Extralvator Abdominoperineal Excision for Advanced Lower Rectal Cancer
Acronym: ELAPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Zhen Jun Wang, Professor, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IELAPE1127
Record Dates: First submitted 2013-11-26; First posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Rectal Cancer
Keywords: Advanced Lower rectal cancer; Extralevator abdominoperineal excision; Circumferential resection margin; Morbidity; Survival
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individual ELAPE (Experimental): Patients will receive Individual ELAPE technique
  Interventions: Procedure: Individual ELAPE
- Conventional ELAPE (Experimental): Patients with advanced lower rectal cancer will receive conventional EALPE technique
  Interventions: Procedure: conventional ELAPE

INTERVENTIONS:
Procedure: conventional ELAPE — device
  Arms: Conventional ELAPE
Procedure: Individual ELAPE — device
  Arms: Individual ELAPE

SUMMARY:
An alternative treatment for low rectal cancer is the extralevator abdominoperineal excision (ELAPE) technique. We aim to compare the outcomes of patients undergoing conventional ELAPE versus Individual ELAPE.

DETAILED DESCRIPTION:
We suppose that the ELAPE technique may be performed according to individual conditions. For the rectal tumors suitable for ELAPE, most of them were circular or nearly circular infiltrating tumors. Patients with these rectal tumors should receive full ELAPE resection. In those rectal tumors not involving the levator ani muscle, the dissection plane may continue close to the external anal sphincter and the levator ani muscle, leaving the ischioanal fat and the terminal branches of the pudendal nerve intact.If the tumor has only penetrated into 1 side of the levator ani muscle, the dissection might include the levator ani muscle and the fat of the ischioanal fossa on the side of the tumor to achieve a clear circumferential resection margin, whereas the ischioanal fat and levator ani muscle on the other side of the tumor may be left

. This individual ELAPE may be as effective as conventional ELAPE while minimizing the operative trauma and the damage to the nerves of the genital organs.

ELIGIBILITY:
Inclusion Criteria:

* Tumor within 5 cm of the anal verge or with a very narrow pelvis
* T3-T4 as determined by preoperative magnetic resonance imaging or endorectal ultrasonography examination or a low tumor is fixed or tethered at rectal examination
* Absence of distant metastases
* Absence of intestinal obstruction

Exclusion Criteria:

* T1-T2 as determined by preoperative magnetic resonance imaging or endorectal ultrasonography examination
* With distant metastases
* With intestinal obstruction
* Pregnancy or lactation
* Allergic constitution to heterogeneous protein
* With operation contraindication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
The perioperative morbidity | three years
  Sexual dysfunction,Urinary retention，Chronic perineal pain，Perineal wound infection，Urinary system infection，Pulmonary infection，Perineal seroma，Peristomal hernia，Abdominal wound infection，Perineal herniation

SECONDARY OUTCOMES:
Three years survival postoperatively | three years

OTHER OUTCOMES:
Three years local recurrence postoperatively | three years

CONTACTS AND LOCATIONS:
Overall Officials: Jiagang Han, Professor, Study Director — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chaoyang Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Han JG, Wang ZJ, Wei GH, Gao ZG, Yang Y, Zhao BC. Randomized clinical trial of conventional versus cylindrical abdominoperineal resection for locally advanced lower rectal cancer. Am J Surg. 2012 Sep;204(3):274-82. doi: 10.1016/j.amjsurg.2012.05.001. PMID 22920402
- See also: Related Info — http://www.ncbi.nlm.nih.gov/m/pubmed/22920402/